CLINICAL TRIAL: NCT01283360
Title: Microbicide Safety and Acceptability in Young Men
Acronym: Project Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1009001; Grant #:1R01HD059533-01A1 (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: High Risk MSM; HIV Negative; 18-30 Years of Age
Keywords: MSM; HIV negative; microbicide; prevention
MeSH Terms: interventions — Tenofovir; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HEC Placebo Gel (Placebo Comparator): In Stage 2, participants will be randomized to receive either tenofovir 1% gel or HEC placebo gel. Following a baseline visit, participants will return to the clinic, where a single dose of the study gel will be administered. Within approximately 30 minutes, rectal swab, stool, and rectal biopsy specimens will be obtained via anoscopy. After a one-week recovery period participants will return to the clinic for assessment. If no significant adverse events (AEs) are reported they will begin to self-administer once-daily outpatient doses of the study gel for 7 days, after which they will return to the clinic for evaluation and specimen collection.
  Interventions: Other: HEC Placebo Gel
- Tenofovir 1% Gel (Active Comparator): In Stage 2, participants will be randomized to receive either tenofovir 1% gel or HEC placebo gel. Following a baseline visit, participants will return to the clinic, where a single dose of the study gel will be administered. Within approximately 30 minutes, rectal swab, stool, and rectal biopsy specimens will be obtained via anoscopy. After a one-week recovery period participants will return to the clinic for assessment. If no significant adverse events (AEs) are reported they will begin to self-administer once-daily outpatient doses of the study gel for 7 days, after which they will return to the clinic for evaluation and specimen collection.
  Interventions: Drug: Tenofovir 1% Gel

INTERVENTIONS:
Other: HEC Placebo Gel — The HEC universal placebo gel for Stage 2 will be supplied by CONRAD (Arlington, VA, USA). Under direction from CONRAD, DPT Laboratories will manufacture the HEC placebo gel and analyze/release the gels under cGMP. DPT Laboratories will fill the applicators with HEC placebo gel to create pre-filled applicators and package each applicator and plunger in a wrapper. Each pre-filled applicator will contain and deliver a dose of approximately 4 mL of HEC gel.
  Arms: HEC Placebo Gel
Drug: Tenofovir 1% Gel — Tenofovir 1% gel will be supplied by CONRAD (Arlington, VA, USA). Under direction from CONRAD, DPT Laboratories will manufacture the tenofovir 1% gel and analyze/release the gels under cGMP. DPT Laboratories will fill the applicators designed for vaginal use with tenofovir 1% gel to create pre-filled applicators and package each applicator and plunger in a wrapper. Each pre-filled applicator will contain and deliver a dose of approximately 4 mL of tenofovir 1% gel (equal to 4.4 g).
  Arms: Tenofovir 1% Gel

SUMMARY:
After completing a screening evaluation, 280 eligible participants, including 40 sex workers, will be enrolled into Stage 1A of the study during which they will undergo a baseline medical evaluation for both history and presence of STIs and anorectal health pathologies or injuries, as well as a detailed Web-based baseline behavioral assessment. The first 140 eligible participants, including 20 sex workers, reporting at least one occasion of unprotected RAI in the previous 3 months will be invited to enroll into Stage 1B. In Stage 1B participants will apply the universal placebo gel (HEC) rectally prior to each episode of RAI over a 3-month period, reporting each use via a phone reporting system; they will complete a Web-based questionnaire and take part in a video teleconference at the end of the 3 months. The first 24 eligible participants completing Stage 1B will be invited to enroll in Stage 2. The subset of sex workers who took part in Stages 1A and 1B will terminate participation at the end of 1B. Eligible participants will be randomized to receive either tenofovir 1% gel or HEC placebo gel as part of Stage 2, the Phase 1 safety study. Following a baseline visit, participants will return to the clinic, where a single dose of the study gel will be administered. Within approximately 30 minutes, rectal swab and rectal biopsy specimens will be obtained via anoscopy. After a one-week recovery period participants will return to the clinic for assessment. If no significant adverse events (AEs) are reported they will begin to self-administer once-daily outpatient doses of the study gel for 7 days, after which they will return to the clinic for evaluation and specimen collection.

DETAILED DESCRIPTION:
Microbicides are products that can be applied in the vagina or rectum to decrease the chances of transmission of sexually transmitted infections (STIs) including HIV. In the US, one of the most vulnerable groups for acquiring HIV infection is young men, especially young Black and Latino men who have sex with men (MSM). This study will be conducted with a young 18-30 year-old ethnically diverse sample of HIV-negative MSM who report engaging in receptive anal intercourse (RAI) using condoms inconsistently or not at all. Our goal is to test whether patterns of use of a placebo rectal gel prior to RAI suggest that the product would be used correctly and consistently in real life circumstances and whether this highly vulnerable population could safely use tenofovir gel, a microbicide candidate. In Version 3.0 of this multicentered protocol, a cohort of 40 male and transgender female sex workers were added to Stages 1A and 1B in order to determine the feasibility of recruitment and retention of men who have sex with men (MSM) with high risk sexual behavior, such as sex workers, for microbicide studies, and their likelihood to use noncondom based HIV prevention strategies. This study will be conducted by the University of Pittsburgh in collaboration with researchers at the HIV Center for Clinical and BehavioralStudies at Columbia University; the Fenway Community Health in Boston; and the University of Puerto Rico Clinical Trial Unit in San Juan, Puerto Rico. Subjects will be enrolled at the University of Pittsburgh, Fenway Community Health, and the University of Puerto Rico. This is a two-stage longitudinal study including a clinical and behavioral evaluation (Stage 1A) with an acceptability and adherence trial (Stage 1B), followed by a Phase 1 randomized, double-blind, multi-site, placebo-controlled trial (Stage 2). Participants who complete Stage 1A are eligible to be selected for enrollment into Stage 1B; a similar transition occurs between Stage 1B and Stage 2.

* In Stage 1A, approximately 280 MSM between the ages of 18-30 will be enrolled, including a subset of 40 sex workers and will undergo a baseline medical evaluation and a detailed Web-based baseline behavioral assessment.
* In Stage 1B, approximately 140 participants from Satge 1A, including a subset of 20 sex workers, will be asked to apply a placebo gel (HEC) rectally prior to each episode of RAI over a 3-month period, reporting each use via a phone reporting system. At the end of the 3 months, participants will complete a Web-based questionnaire and take part in a video teleconference.The first 42 eligible participants, excluding the mal and transgender female sex worker cohort, (approximately 14 at each site) completing Stage 1B with a reported adherence of 80% or greater will be invited to enroll in Stage 2.
* In Stage 2, approximately 24 eligible participants from Stage 1B will progress to Stage 2 and be randomized at a 1:1 ratio to tenofovir 1% gel or HEC placebo gel.Following a baseline visit, participants will return to the clinic, where a single dose of the study gel will be administered. Within approximately 30 minutes, rectal swab, stool, and rectal biopsy specimens will be obtained via anoscopy. After a one-week recovery period participants will return to the clinic for assessment. If no significant adverse events(AEs) are reported they will begin to self-administer once-daily outpatient doses of the study gel for 7 days, after which they will return to the clinic for evaluation and specimen collection.

ELIGIBILITY:
Inclusion Criteria for Participants in Stage 1A (non sex-workers):

1. Willing and able to provide written informed consent to take part in the study
2. Willing and able to communicate in English or Spanish
3. Must agree not to participate in other drug trials
4. Biologically male and identifies as male
5. Age 18-30 years at screening
6. HIV-1 status antibody negative or unknown per patient report
7. Understands and agrees to local STI reporting requirements
8. Able and willing to provide adequate information for locator purposes
9. Availability to return for all study visits, barring unforeseen circumstances
10. A history of consensual RAI at least once in past month
11. Reporting at least one occasion of unprotected RAI in the prior year* In order to identify participants at increased risk for acquiring HIV

Inclusion Criteria for Participants in Stage 1A (sex-workers):

1. Willing and able to provide written informed consent to take part in the study
2. Willing and able to communicate in English or Spanish
3. Must agree not to participate in other drug trials
4. Biologically male, including male-to-female transgender women
5. Age 18-30 years at screening
6. HIV-1 status antibody negative or unknown per patient report
7. Understands and agrees to local STI reporting requirements
8. Able and willing to provide adequate information for locator purposes
9. Availability to return for all study visits, barring unforeseen circumstances
10. A history of consensual RAI at least once in past month
11. Reporting at least one occasion of unprotected RAI in the prior year*
12. Reporting at least two occasions of RAI as part of transactional sex (i.e., having received money or other goods/services in exchange for sex) in the prior 2 months*

    * In order to identify participants at increased risk for acquiring HIV

Inclusion Criteria for Participants in Stage 1B (both sex workers and non sex-workers):

1. Completed Stage 1A
2. HIV-1 uninfected at screening based on HIV rapid test results
3. Reports unprotected RAI in the prior three months on at least one occasion* In order to obtain acceptability data from individuals most likely to benefit from microbicide availability
4. Availability to return for all Stage 1B visits, barring unforeseen circumstances

Inclusion Criteria for Participants in Stage 2:

1. Completed study stage 1AB
2. HIV-1 uninfected at screening based on HIV rapid test results
3. Availability to return for all Stage 2 visits, barring unforeseen circumstances

Exclusion Criteria for Participants in Stage 1A (both sex workers and non sex-workers):

1. Any condition or prior therapy that, in the opinion of the investigator, would make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease

Exclusion Criteria for Participants in Stage 1B (both sex workers and non sex-workers):

1. Clinical or laboratory diagnosis of active rectal infection requiring treatment per current CDC guidelines. Infections requiring treatment include Chlamydia (CT), gonorrhea (GC), syphilis, active HSV lesions, chancroid, genital sores or ulcers, and if clinically indicated, genital warts. Note that an HSV-2 seropositive diagnosis with no active lesions is allowed, since treatment is not required
2. Positive Hepatitis B surface antigen test indicating hepatitis B infection
3. Allergy to methylparaben, propylparaben, or latex
4. History of significant drug allergy or recurrent urticaria
5. History of inflammatory bowel disease
6. Currently engage or plan to engage in unprotected RAI with HIV-infected partners
7. By participant report planning to receive another investigational drug while participating in this study
8. Any other condition or prior therapy that, in the opinion of the investigator, would make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease

Exclusion Criteria for Participants in Stage 2:

1. Meet any of the exclusion criteria for Stage 1B
2. Reporting a history of transactional sex (i.e., having received money or other goods/services in exchange for sex) in the prior 6 months
3. Undergoing or completed gender reassignment
4. Grade 2 or higher liver function, creatinine, coagulation, electrolyte, or hematology abnormality in accordance with DAIDS toxicity table values (normal values based on site specific laboratory criteria) at screening (or Visit 2 PT/INR for coagulation), and confirmed by retest/and or redraw
5. History of significant gastrointestinal bleeding
6. History of inflammatory bowel disease
7. Abnormalities of the rectal mucosa, or significant rectal symptom(s), which in the opinion of the clinician represents a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids
8. Per participant report, anticipated use and/or unwillingness to abstain from the following medications during the period of Stage 2 study participation:

   1. Heparin, including Lovenox®
   2. Warfarin
   3. Plavix® (clopidogrel bisulfate)
   4. Aspirin >81 mg per day
   5. Non-steroidal anti-inflammatory drugs (NSAIDS)
   6. Any other drugs that are associated with increased likelihood of bleeding following rectal biopsy
9. By participant report, use of systemic immunomodulatory medications within the 4 weeks prior to the Stage 2 Enrollment Visit and throughout study participation
10. By participant report, use of rectally administered medications, rectally administered products (including condoms) containing N-9, or any investigational products within the 2 weeks or 10 half-lives of the drug, whichever is longer, prior to the Stage 2 Enrollment Visit, or is planning to receive another investigational drug while participating in this study
11. Any other condition or prior therapy that, in the opinion of the investigator, would make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease -

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 249 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Stage 1AB Primary behavioral outcomes | 3 months
  * Identification of factors related to acceptability and adherence
  * Proportion of participants who report via the acceptability questionnaire that they would be very likely to use a similar candidate microbicide gel during receptive anal intercourse (RAI)
  * Proportion of RAI episodes in which the gel was used
  * Comparison between self-reports of placebo gel use and applicator counts in Stage 1B
Stage 1AB Primary clinical outcome | 3 months
  the presence of STIs and anal and rectal pathologies as detected by standard anoscopy
Stage 2 Primary clinical outcomes | 6 months
  Grade 2 or higher AEs, as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 and/or Addenda 3 (Rectal Grading Tables for Use in Microbicide Studies).
Stage 2 Behavioral | 6 months
  * Identification of factors related to acceptability and adherence
  * Proportion of participants who report via the acceptability questionnaire that they would be very likely to use a similar candidate microbicide gel during receptive anal intercourse (RAI)
  * Proportion of RAI episodes in which the gel was used by participants
  * Comparison between self-reports of gel use and applicator counts

SECONDARY OUTCOMES:
Stage 1AB Secondary clinical endpoint | 3 months
  Percent of agreement between reports of anal and rectal pathologies by two assessment methods (standard anoscopy versus high-resolutions anoscopy).
Stage 2 Secondary behavioral outcomes | 6 months
  * Identification of factors related to sexual behaviors (e.g., douching, lubricant use, recreational drug use, condom use, partner selection)
  * Prevalence of risky sexual practices, douching, lubricant use, recreational drug use, and condom use
Stage 1AB Secondary behavioral outcomes | 3 months
  * Identification of factors related to sexual behaviors (e.g., condom use, lubricant use, douching, risky sexual practices, and recreational drug use)
  * Prevalence of condom use, lubricant use, douching, risky sexual practices, and recreational drug use
Stage 2 Behavioral | 6 months
  * Identification of factors related to sexual behaviors (e.g., douching, lubricant use, recreational drug use, condom use, partner selection)
  * Prevalence of risky sexual practices, douching, lubricant use, recreational drug use, and condom use

OTHER OUTCOMES:
Stage 1AB Tertiary Behavioral | 3 months
  * Proportion of individuals identifying as sex workers screened to individuals enrolled in the sex worker cohort
  * Proportion of visits completed by participants enrolled in the sex worker cohort
  * Likelihood of using microbicide gels, PrEP, or a rapid HIV Home Test with clients and non-commercial partners for individuals identifying as sex workers

CONTACTS AND LOCATIONS:
Overall Officials: Ian McGowan, MD, PhD, Principal Investigator — University of Pittsburgh; Alex Carballo-Dieguez, PhD, Principal Investigator — New York State Psychiatric Institute and Columbia University; Lynne M. Mofensen, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (3):
- United States (2):
  - The Fenway Institute-Fenway Community Health, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- University of Puerto Rico Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Derived] McGowan I, Cranston RD, Mayer KH, Febo I, Duffill K, Siegel A, Engstrom JC, Nikiforov A, Park SY, Brand RM, Jacobson C, Giguere R, Dolezal C, Frasca T, Leu CS, Schwartz JL, Carballo-Dieguez A. Project Gel a Randomized Rectal Microbicide Safety and Acceptability Study in Young Men and Transgender Women. PLoS One. 2016 Jun 30;11(6):e0158310. doi: 10.1371/journal.pone.0158310. eCollection 2016. PMID 27362788